CLINICAL TRIAL: NCT00492284
Title: A Multicenter, Randomized, Single-masked Study Comparing Reduced-fluence Visudyne®-Lucentis® Combination Therapies and Lucentis® Monotherapy in Subjects With Choroidal Neovascularization (CNV) Secondary to AMD.
Brief Title: Reduced Fluence Visudyne-Anti-VEGF-Dexamethasone In Combination for AMD Lesions (RADICAL)
Acronym: RADICAL
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: QLT Inc. (Industry)
Responsible Party: Dr. Oscar Cuzzani, QLT Inc.
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BPD OCR 022
Record Dates: First submitted 2007-06-25; First posted 2007-06-27 (Estimated); Results first posted 2010-06-22 (Estimated); Last update posted 2011-06-02 (Estimated); Status verified 2011-05

CONDITIONS: Choroidal Neovascularization; Macular Degeneration
Keywords: Macular Degeneration; AMD; CNV; Choroidal neovascularization; Photodynamic therapy; CNV Secondary to Age Related Macular Degeneration
MeSH Terms: conditions — Choroidal Neovascularization; Macular Degeneration | interventions — Verteporfin; Photochemotherapy; Ranibizumab; Dexamethasone

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1/4 Fluence Triple Therapy (Experimental): Very low fluence Visudyne followed by intravitreal Lucentis-Dexamethasone triple therapy [within 2 hours] administered on Day 0, and then as required every 2 months thereafter
  Interventions: Drug: verteporfin; Drug: ranibizumab; Drug: dexamethasone
- 1/2 Fluence Triple Therapy (Experimental): Reduced-fluence Visudyne followed by intravitreal Lucentis-Dexamethasone triple therapy [within 2 hours] administered on Day 0, and then as required every 2 months thereafter
  Interventions: Drug: verteporfin; Drug: ranibizumab; Drug: dexamethasone
- 1/2 Fluence Double Therapy (Experimental): Reduced-fluence Visudyne followed by Lucentis double therapy [within 2 hours] administered on Day 0, and then as required every 2 months thereafter
  Interventions: Drug: verteporfin; Drug: ranibizumab
- Ranibizumab (Experimental): Lucentis monotherapy administered on Day 0, Month 1 and Month 2, and then as required monthly thereafter
  Interventions: Drug: ranibizumab

INTERVENTIONS:
Drug: verteporfin — Reduced-fluence Visudyne (25 J/cm2, 300 mW/cm2, 83 seconds)
  Other Names: Visudyne; photodynamic therapy
  Arms: 1/2 Fluence Double Therapy; 1/2 Fluence Triple Therapy
Drug: verteporfin — Very-low fluence Visudyne (15 J/cm2, 180 mW/cm2, 83 seconds)
  Other Names: Visudyne; photodynamic therapy
  Arms: 1/4 Fluence Triple Therapy
Drug: ranibizumab — 0.5 mg intravitreal injection
  Other Names: Lucentis
Drug: dexamethasone — 0.5 mg intravitreal injection
  Arms: 1/2 Fluence Triple Therapy; 1/4 Fluence Triple Therapy

SUMMARY:
The objective of this study is to determine if combination therapy (reduced-fluence Visudyne followed by Lucentis [within 2 hours] or either of two regimens of reduced-fluence Visudyne followed by Lucentis-Dexamethasone triple therapy [within 2 hours]) reduces retreatment rates compared with Lucentis monotherapy while maintaining similar vision outcomes and an acceptable safety profile.

ELIGIBILITY:
Inclusion Criteria:

* Treatment naive for choroidal neovascularization (CNV) secondary to age-related macular degeneration (AMD) in the study eye except for laser treatment outside the subfoveal area
* Subfoveal CNV due to AMD
* CNV must be = or >50 % of the entire lesion
* All lesion composition types with a lesion greatest linear dimension (GLD) < 5400 microns (approximately = or <9 disc areas [DA])
* Best-corrected Early Treatment Diabetic Retinopathy Study (ETDRS) visual acuity (VA score) of 25 - 73 letters (approximate Snellen equivalent of 20/40 - 20/320), inclusive

Exclusion Criteria:

* Subfoveal geographic atrophy or subfoveal fibrosis of the study eye
* Intraocular surgery within 3 months of enrollment
* Inability to attend the protocol-required visits
* Known allergies or hypersensitivity to any of the study treatments.
* Other systemic diseases or active uncontrolled infections that would make subject a poor medical risk
* Uncontrolled glaucoma, defined as (1)subject is on >1 glaucoma medication (includes combination treatments) or (2)subject has glaucoma that could lead to progressive visual field deterioration
* If subject has had a stroke within the last year

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 162 (Actual)
Dates: Start 2007-07; Primary Completion 2009-05 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Henry Hudson, MD, Principal Investigator — Retina Centers, PC; Allen Ho, MD, Principal Investigator — Retina Diagnostic & Treatment Associates, LLC; Andrew Strong, Ph.D, Study Chair — QLT Inc.; Oscar Cuzzani, MD, Study Director — QLT Inc.
Locations (26):
- United States (21):
  - Mobile, Alabama
  - Phoenix, Arizona
  - Retina Centers, PC, Tucson, Arizona
  - Beverly Hills, California
  - Campbell, California
  - Los Angeles, California
  - Poway, California
  - Sacramento, California
  - Torrance, California
  - Fort Myers, Florida
  - Indianapolis, Indiana
  - Davenport, Iowa
  - Missoula, Montana
  - Omaha, Nebraska
  - Portsmouth, New Hampshire
  - Portland, Oregon
  - Philadelphia, Pennsylvania
  - West Mifflin, Pennsylvania
  - Arlington, Texas
  - Temple, Texas
  - Seattle, Washington
- Canada (5):
  - Calgary, Alberta
  - Vancouver, British Columbia
  - Halifax, Nova Scotia
  - London, Ontario
  - Toronto, Ontario

RESULTS

PARTICIPANT FLOW:
Groups:
- 1/4 Fluence Triple Therapy: Very low fluence Visudyne (15 J/cm2: 180 mW/cm2 for 83 seconds) followed by intravitreal Lucentis (0.5 mg)-Dexamethasone (0.5 mg) triple therapy [within 2 hours] on Day 0 and then as required every 2 months thereafter
- 1/2 Fluence Triple Therapy: Reduced-fluence Visudyne (25 J/cm2: 300 mW/cm2 for 83 seconds) followed by intravitreal Lucentis (0.5 mg)-Dexamethasone (0.5 mg) triple therapy [within 2 hours] on Day 0 and then as required every 2 months thereafter
- 1/2 Fluence Double Therapy: Reduced-fluence Visudyne (25 J/cm2: 300 mW/cm2 for 83 seconds) followed by intravitreal Lucentis (0.5 mg) double therapy [within 2 hours]
- Ranibizumab: Lucentis monotherapy (0.5 mg)on Day 0, Month 1, and Month 2, and then as required monthly thereafter
Period: Overall Study
Arm/Group | 1/4 Fluence Triple Therapy | 1/2 Fluence Triple Therapy | 1/2 Fluence Double Therapy | Ranibizumab
Started | 39 | 39 | 43 | 41
Completed | 38 | 35 | 37 | 31
Not Completed | 1 | 4 | 6 | 10
Not completed — Adverse Event | 0 | 1 | 1 | 2
Not completed — Lost to Follow-up | 0 | 0 | 3 | 1
Not completed — Death | 0 | 3 | 2 | 5
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 1/4 Fluence Triple Therapy | 1/2 Fluence Triple Therapy | 1/2 Fluence Double Therapy | Ranibizumab | Total
Number analyzed (Participants) | 39 | 39 | 43 | 41 | 162
Age Continuous [Mean (Standard Deviation); unit: years] | 78 (8) | 78 (8) | 79 (6) | 79 (5) | 79 (7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 24 | 23 | 28 | 95
  Male | 19 | 15 | 20 | 13 | 67
Lesion composition [Number; unit: participants]
  Minimally classic | 6 | 4 | 9 | 8 | 27
  Occult no classic | 10 | 16 | 20 | 18 | 64
  Predominantly classic | 23 | 19 | 14 | 15 | 71
Central retinal thickness [Mean (Standard Deviation); unit: micron] | 318.3 (95.9) | 337.3 (106.8) | 337.3 (121.4) | 311.9 (95.5) | 326.3 (105.4)
Lesion size (greatest linear dimension) [Mean (Standard Deviation); unit: micron] | 2778.8 (1025.6) | 2740.1 (846.1) | 2796.1 (1122.8) | 3118.4 (1155.7) | 2860.1 (1049.4)
Study Eye Best-corrected Visual Acuity Score (ETDRS chart) [Mean (Standard Deviation); unit: Letters read on ETDRS chart] — Early Treatment Diabetic Retinopathy Study (ETDRS) method at 4 meters. Worst = 0; best = 100
  Letters read on ETDRS chart | 58.1 (11.8) | 55.6 (11.2) | 53.3 (11.9) | 56.0 (13.1) | 55.7 (12.0)

OUTCOME MEASURES:

1. Primary Outcome: Mean Number of Retreatments (Day 0 Excluded)
Description: Retreatment was defined in the protocol as study treatment administered after Day 0. For the analyses of retreatment, any study treatment that was administered was considered to be a retreatment, and combination therapy was considered to be one retreatment, even though two or three treatment procedures were done. In the combination therapy groups, if a ranibizumab injection was given because retreatment was indicated and the previous combination treatment was less than 2 months before, the ranibizumab injection was counted as a retreatment.
Time Frame: Month 1 to Month 12
Population: Intent-to-treat
Measure: Mean (95% Confidence Interval); unit: number of retreatments
Arm/Group | 1/4 Fluence Triple Therapy | 1/2 Fluence Triple Therapy | 1/2 Fluence Double Therapy | Ranibizumab
Number analyzed (Participants) | 39 | 39 | 43 | 41
number of retreatments | 3.97 (3.12) [2.96 to 4.98] | 3.00 (2.55) [2.17 to 3.83] | 4.05 (2.93) [3.15 to 4.95] | 5.39 (2.97) [4.45 to 6.33]

2. Primary Outcome: Mean Change From Baseline in Study Eye Best-corrected VA Score (ETDRS Chart)
Description: Early Treatment Diabetic Retinopathy Study (ETDRS) method at 4 meters. Worst = 0; best = 100
Time Frame: Baseline to Month 12
Population: Intent-to-treat and last observation carried forward
Measure: Mean (95% Confidence Interval); unit: Letters read on ETDRS chart
Arm/Group | 1/4 Fluence Triple Therapy | 1/2 Fluence Triple Therapy | 1/2 Fluence Double Therapy | Ranibizumab
Number analyzed (Participants) | 39 | 39 | 43 | 41
Letters read on ETDRS chart | 3.6 (13.8) [-0.9 to 8.1] | 6.8 (13.4) [2.4 to 11.1] | 5.0 (14.2) [0.6 to 9.3] | 6.5 (15.5) [1.7 to 11.4]

3. Secondary Outcome: Mean Number of Retreatments (Day 0 Excluded)
Description: as for outcome 1
Time Frame: Month 1 to Month 24
Population: Intent-to-treat
Measure: Mean (95% Confidence Interval); unit: number of retreatments
Arm/Group | 1/4 Fluence Triple Therapy | 1/2 Fluence Triple Therapy | 1/2 Fluence Double Therapy | Ranibizumab
Number analyzed (Participants) | 39 | 39 | 43 | 41
number of retreatments | 5.92 [4.35 to 7.49] | 4.34 [3.09 to 5.60] | 5.92 [4.46 to 7.38] | 8.68 [6.74 to 10.62]

4. Secondary Outcome: Mean Change From Baseline in Study Eye Best-Corrected VA Score
Description: Early Treatment Diabetic Retinopathy Study (ETDRS) method at 4 meters. Worst = 0; best = 100
Time Frame: Baseline to Month 24
Measure: Mean (95% Confidence Interval); unit: Letters read on ETDRS chart
Arm/Group | 1/4 Fluence Triple Therapy | 1/2 Fluence Triple Therapy | 1/2 Fluence Double Therapy | Ranibizumab
Number analyzed (Participants) | 39 | 39 | 43 | 41
Letters read on ETDRS chart | -0.2 [-5.7 to 5.4] | 1.1 [-4.3 to 6.4] | -0.3 [-6.2 to 5.6] | 4.4 [-1.5 to 10.2]

5. Secondary Outcome: Percentage of Subjects With >=15 Letters of Visual Acuity Gained From Baseline
Time Frame: Baseline to Month 12, Baseline to Month 24
Population: Intent-to-treat and last observation carried forward
Measure: Mean (95% Confidence Interval); unit: Percentage of participants
Arm/Group | 1/4 Fluence Triple Therapy | 1/2 Fluence Triple Therapy | 1/2 Fluence Double Therapy | Ranibizumab
Number analyzed (Participants) | 39 | 39 | 43 | 41
Percentage of participants
  Baseline to Month 12 | 25.6 [11.9 to 39.3] | 30.8 [16.3 to 45.3] | 25.6 [12.5 to 38.6] | 24.4 [11.2 to 37.5]
  Baseline to Month 24 | 20.5 [7.8 to 33.2] | 15.4 [4.1 to 26.7] | 16.3 [5.2 to 27.3] | 26.8 [13.3 to 40.4]

6. Secondary Outcome: Percentage of Subjects With >=0 Letter Gain of Visual Acuity From Baseline
Time Frame: Baseline to Month 12, Baseline to Month 24
Population: Intent-to-treat and last observation carried forward
Measure: Mean (95% Confidence Interval); unit: Percentage of participants
Arm/Group | 1/4 Fluence Triple Therapy | 1/2 Fluence Triple Therapy | 1/2 Fluence Double Therapy | Ranibizumab
Number analyzed (Participants) | 39 | 39 | 43 | 41
Percentage of participants
  Baseline to Month 12 | 64.1 [49.0 to 79.2] | 82.1 [70.0 to 94.1] | 69.8 [56.0 to 83.5] | 70.7 [56.8 to 84.7]
  Baseline to Month 24 | 61.5 [46.3 to 76.8] | 66.7 [51.9 to 81.5] | 60.5 [45.9 to 75.1] | 70.7 [56.8 to 84.7]

7. Secondary Outcome: Percentage of Subjects With >=15 Letters of Visual Acuity Lost From Baseline
Time Frame: Baseline to Month 12, Baseline to Month 24
Population: Intent-to-treat and last observation carried forward
Measure: Mean (95% Confidence Interval); unit: Percentage of participants
Arm/Group | 1/4 Fluence Triple Therapy | 1/2 Fluence Triple Therapy | 1/2 Fluence Double Therapy | Ranibizumab
Number analyzed (Participants) | 39 | 39 | 43 | 41
Percentage of participants
  Baseline to Month 12 | 12.8 [2.3 to 23.3] | 7.7 [0 to 16.1] | 11.6 [2.0 to 21.2] | 7.3 [0 to 15.3]
  Baseline to Month 24 | 20.5 [7.8 to 33.2] | 15.4 [4.1 to 26.7] | 20.9 [8.8 to 33.1] | 14.6 [3.8 to 25.5]

8. Secondary Outcome: Mean Change From Baseline in Central Retinal Thickness
Time Frame: Baseline to Month 12, Baseline to Month 24
Population: Intent-to-treat and last observation carried forward
Measure: Mean (Standard Deviation); unit: micron
Arm/Group | 1/4 Fluence Triple Therapy | 1/2 Fluence Triple Therapy | 1/2 Fluence Double Therapy | Ranibizumab
Number analyzed (Participants) | 39 | 39 | 43 | 41
micron
  Baseline to Month 12 | -115.9 (97.4) | -122.2 (104.8) | -137.8 (122.3) | -100.3 (90.1)
  Baseline to Month 24 | -110.2 (93.6) | -123.9 (97.1) | -121.0 (126.6) | -103.1 (99.1)

9. Secondary Outcome: Mean Change From Baseline in Lesion Size
Description: Mean change from baseline in lesion size measured as greatest linear dimension (GLD) of the lesion
Time Frame: Baseline to Month 12, Baseline to Month 24
Population: Intent-to-treat and last observation carried forward
Measure: Mean (Standard Deviation); unit: micron
Arm/Group | 1/4 Fluence Triple Therapy | 1/2 Fluence Triple Therapy | 1/2 Fluence Double Therapy | Ranibizumab
Number analyzed (Participants) | 39 | 39 | 43 | 41
micron
  Baseline to Month 12 | 77.2 (960.3) | -20.4 (1550.7) | 152.0 (1415.5) | -192.6 (672.5)
  Baseline to Month 24 | 94.8 (865.1) | -103.3 (1326.1) | -112.5 (1209.4) | -205.3 (653.4)

ADVERSE EVENTS:
Time Frame: Month 0 to Month 24/last visit
Arm/Group | 1/4 Fluence Triple Therapy | 1/2 Fluence Triple Therapy | 1/2 Fluence Double Therapy | Ranibizumab
Serious Adverse Events (participants affected / at risk) | 10/39 | 13/39 | 15/43 | 19/41
Other Adverse Events (participants affected / at risk) | 36/39 | 36/39 | 36/43 | 37/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1/4 Fluence Triple Therapy (N=39) | 1/2 Fluence Triple Therapy (N=39) | 1/2 Fluence Double Therapy (N=43) | Ranibizumab (N=41)
AV block complete (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
AV block second degree (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal Pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Accidental Injury (General disorders) | 0 (0) | 2 (2) | 1 (1) | 1 (1)
Acute kidney failure (Renal and urinary disorders) | 0 (0) | 2 (3) | 0 (0) | 2 (2)
Anaphylactoid Reaction (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Angina pectoris (Cardiac disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Aplastic anemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arrhythmia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Arteriosclerosis (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Aspiration pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Breast carcinoma (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Bundle Branch Block (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cardiovascular disorder (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Cellulitis (General disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Cerebral infarct (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Chest pain (General disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Cholecystitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cholelithiasis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Congestive Heart Failure (Cardiac disorders) | 0 (0) | 2 (2) | 1 (1) | 3 (3)
Death (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Diabetes Mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Endocarditis (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal carcinoma (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Gastrointestinal neoplasia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Healing abnormal (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Heart arrest (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hernia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Hypotension (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypoxia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Increased intraocular pressure (study eye) (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infection (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Infection bacterial (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intestinal perforation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Kidney failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lung edema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neck pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pathological Fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3) | 0 (0) | 3 (3)
Postural Hypotension (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Psychosis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pyogenic arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Retinal detachment (study eye) (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Retinal tear (study eye) (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sepsis (General disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Syncope (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Thinking abnormal (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Vascular anomaly (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vertigo (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Viral infection (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vision decreased (study eye) (Eye disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Visual field defect (study eye) (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vitreous hemorrhage (study eye) (Eye disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Cardiomyopathy (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Coronary artery disorder (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Peripheral vascular disorder (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pulmonary embolus (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cholangitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Liver damage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Adrenal disorder (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood dyscrasia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypomagnesemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bone neoplasm (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Confusion (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Convulsion (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Apnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5.0% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | 1/4 Fluence Triple Therapy (N=39) | 1/2 Fluence Triple Therapy (N=39) | 1/2 Fluence Double Therapy (N=43) | Ranibizumab (N=41)
Accidental Injury (General disorders) | 6 (11) | 5 (9) | 7 (11) | 9 (15)
Age-related Macular Degeneration progression (fellow eye) (Eye disorders) | 3 (3) | 8 (8) | 1 (1) | 2 (2)
Anemia (Blood and lymphatic system disorders) | 2 (2) | 3 (3) | 2 (2) | 2 (2)
Anxiety (Nervous system disorders) | 3 (3) | 0 (0) | 2 (2) | 3 (3)
Asthenia (General disorders) | 1 (1) | 4 (5) | 5 (7) | 3 (3)
Back pain (General disorders) | 4 (4) | 2 (2) | 0 (0) | 1 (1)
Blepharitis (fellow eye) (Eye disorders) | 0 (0) | 4 (4) | 0 (0) | 0 (0)
Blepharitis (study eye) (Eye disorders) | 0 (0) | 4 (4) | 1 (1) | 1 (1)
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 4 (4) | 2 (2) | 3 (3)
Cataract (fellow eye) (Eye disorders) | 2 (2) | 4 (4) | 2 (2) | 4 (4)
Cataract (study eye) (Eye disorders) | 2 (2) | 4 (4) | 6 (6) | 1 (1)
Chest pain (General disorders) | 2 (2) | 1 (1) | 2 (2) | 1/1 (1)
Cholelithiasis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
Conjunctivitis (study eye) (Eye disorders) | 2 (4) | 3 (3) | 2 (2) | 2 (2)
Corneal lesion (study eye) (Eye disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Cough increased (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 6 (6) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 4 (4) | 2 (2) | 2 (2)
Dizziness (Nervous system disorders) | 4 (4) | 5 (5) | 1 (1) | 1 (1)
Ecchymosis (Blood and lymphatic system disorders) | 1 (1) | 3 (3) | 2 (3) | 2 (5)
Eye itching (fellow eye) (Eye disorders) | 1 (1) | 3 (3) | 0 (0) | 3 (3)
Eye itching (study eye) (Eye disorders) | 2 (2) | 3 (3) | 1 (1) | 3 (4)
Eye pain (study eye) (Eye disorders) | 7 (15) | 9 (11) | 9 (15) | 10 (23)
Flu syndrome (General disorders) | 1 (1) | 2 (2) | 0 (0) | 4 (4)
Headache (General disorders) | 3 (4) | 1 (2) | 4 (4) | 2 (2)
Hypercholesterolemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 3 (3) | 2 (2)
Hyperlipemia (Metabolism and nutrition disorders) | 0 (0) | 3 (3) | 1 (1) | 2 (2)
Hypertension (Cardiac disorders) | 7 (9) | 2 (2) | 7 (7) | 5 (5)
Increased intraocular pressure (study eye) (Eye disorders) | 4 (4) | 4 (12) | 6 (8) | 6 (8)
Infection (General disorders) | 7 (9) | 7 (9) | 5 (8) | 8 (10)
Infusion-related back pain (General disorders) | 1 (1) | 2 (5) | 4 (8) | 0 (0)
Injection site pain (General disorders) | 1 (1) | 1 (1) | 3 (4) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 3 (3) | 4 (4) | 3 (3)
Pain (General disorders) | 3 (3) | 4 (4) | 4 (4) | 5 (5)
Peripheral edema (Metabolism and nutrition disorders) | 0 (0) | 3 (3) | 2 (2) | 2 (2)
Peripheral vascular disorder (Cardiac disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 3 (3) | 0 (0) | 3 (3)
Syncope (Cardiac disorders) | 1 (1) | 5 (5) | 2 (2) | 0 (0)
Urinary tract infection (Renal and urinary disorders) | 2 (8) | 3 (3) | 4 (4) | 6 (8)
Vision abnormal (study eye) (Eye disorders) | 8 (10) | 1 (1) | 7 (10) | 4 (4)
Vision decreased (study eye) (Eye disorders) | 5 (6) | 4 (4) | 6 (8) | 1 (1)
Visual field defect (study eye) (Eye disorders) | 5 (5) | 0 (0) | 2 (2) | 4 (4)
Vitreous disorder (study eye) (Eye disorders) | 4 (4) | 2 (2) | 3 (3) | 5 (5)
Abdominal pain (General disorders) | 1 (1) | 1 (1) | 2 (2) | 2 (2)
Allergic reaction (General disorders) | 2 (2) | 2 (2) | 1 (1) | 3 (3)
Injection site extravasation (General disorders) | 2 (2) | 1 (1) | 3 (3) | 0 (0)
Bradycardia (Cardiac disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Cardiovascular disorder (Cardiac disorders) | 2 (3) | 0 (0) | 2 (5) | 1 (1)
Cerebral ischemia (Cardiac disorders) | 1 (1) | 3 (3) | 0 (0) | 1 (1)
Hemorrhage (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Vascular anomaly (Cardiac disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 3 (3) | 1 (1) | 2 (2) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 2 (2) | 2 (2) | 1 (2)
Dyspepsia (Gastrointestinal disorders) | 2 (3) | 0 (0) | 1 (2) | 1 (1)
Gastrointestinal disorder (Gastrointestinal disorders) | 1 (1) | 1 (1) | 4 (4) | 2 (2)
Periodontal abscess (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1) | 2 (3)
Hypothyroidism (Gastrointestinal disorders) | 2 (2) | 3 (3) | 0 (0) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 4 (4) | 4 (4) | 2 (2) | 1 (1)
Bone disorder (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 0 (0) | 1 (1)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 4 (4) | 3 (3) | 1 (1)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 2 (2) | 0 (0)
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (2) | 0 (0) | 0 (0)
Acute brain syndrome (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Dementia (Nervous system disorders) | 2 (2) | 2 (2) | 1 (1) | 1 (1)
Depression (Nervous system disorders) | 2 (2) | 1 (1) | 1 (1) | 1 (1)
Neuralgia (Nervous system disorders) | 2 (3) | 1 (1) | 0 (0) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 0 (0) | 2 (2)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 4 (4) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 1 (1) | 1 (1)
Skin carcinoma (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2) | 1 (1) | 2 (2)
Skin disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 3 (4)
Conjunctivitis (fellow eye) (Eye disorders) | 2 (3) | 1 (1) | 0 (0) | 0 (0)
Dry eyes (fellow eye) (Eye disorders) | 2 (2) | 0 (0) | 1 (1) | 1 (1)
Retinal disorder (fellow eye) (Eye disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Vitreous detachment (fellow eye) (Eye disorders) | 1 (1) | 1 (1) | 0 (0) | 3 (3)
Diplopia (study eye) (Eye disorders) | 0 (0) | 3 (3) | 1 (1) | 1 (1)
Dry eyes (study eye) (Eye disorders) | 3 (3) | 1 (2) | 1 (1) | 1 (1)
Retinal disorder (study eye) (Eye disorders) | 3 (3) | 4 (5) | 1 (1) | 1 (1)
Subconjunctival hemorrhage (study eye) (Eye disorders) | 2 (2) | 2 (4) | 0 (0) | 2 (2)
Cystitis (Renal and urinary disorders) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Kidney function abnormal (Renal and urinary disorders) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Prostatic disorder (Renal and urinary disorders) | 1 (1) | 2 (2) | 2 (3) | 2 (2)

LIMITATIONS AND CAVEATS:
Retreatment and vision analysis limitations, sample size, lack of standard monotherapy regimen used in practice, no treatment regimen approved by regulatory authorities, potential for bias in FA assessment, no central reading center, single-masked

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Publication materials will be reviewed and commented on by the Sponsor prior to submission for publication; Names of all Investigators and Sponsor representatives responsible for study design and analysis of results will be disclosed in the publication.